CLINICAL TRIAL: NCT00430651
Title: Multicenter Randomized Phase III Study Comparing Docetaxel With Carboplatin Versus Docetaxel Single Agent as Second Line Treatment in Patients With Non-Small Cell Lung Cancer (NSCLC).
Brief Title: Docetaxel and Carboplatin Versus Docetaxel as Second Line Treatment in Patients With Non-Small-Cell Lung Carcinoma (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: V.Georgoulias, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/04.14
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; 2nd line chemotherapy; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Carboplatin

ARMS (2):
- 1 (Experimental): Docetaxel + Carboplatin
  Interventions: Drug: Docetaxel; Drug: Carboplatin
- 2 (Experimental): Docetaxel
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50 mg/m2 IV on days 1 and 15 every 28 days for 6 cycles
  Other Names: Taxotere
Drug: Carboplatin — Docetaxel 50 mg/m2 IV over 1 hour followed by Carboplatin 4 AUC IV over 1 hour on days 1 and 15
  Arms: 1

SUMMARY:
This trial will compare the effectiveness of Docetaxel with or without Carboplatin as second line chemotherapy in patients with Non-Small Cell Lung Cancer, who have not been treated previously with Docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC.
* ECOG Performance Status 0-2.
* No previous treatment with Docetaxel.
* Measurable Disease.
* Brain metastases that have been treated with radiotherapy should be stable and asymptomatic.
* Adequate liver kidney and bone marrow function.
* Patients must be able to understand the nature of this study and give written informed consent.

Exclusion Criteria:

* Active cardiac disease: unstable angina or onset of angina within last 3 months, myocardial infarction within 6 months, congestive heart failure > class II, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Women who are pregnant or lactating.
* Unknown HIV, chronic hepatitis B or chronic hepatitis C infections.
* Serious neurologic or psychiatric disease.
* Second primary malignancy within the past 5 years, except nonmelanomas skin cancer or in situ carcinoma of the cervix.
* Active uncontrolled infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2004-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the overall survival between the two treatment groups | 1 year

SECONDARY OUTCOMES:
Comparison of the objective response rates between the two treatment groups | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Evaluation and comparison of the toxicity between the two treatment groups | Toxicity assessment on each chemotherapy cycle
Measurement and comparison of the health-related quality of life of patients on both treatment groups | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (10):
- Greece (10):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athnes, Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Sotiria" General Hospital, 1st, 3rd, 6th, 7th, 8th Dep of Pulmonary Diseases, Athens
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - "Metaxa's" Anticancer Hospital of Pireaus, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki